CLINICAL TRIAL: NCT04719143
Title: Effects of Insomnia Treatment on Metabolism in Patients With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 831841
Record Dates: First submitted 2020-12-09; First posted 2021-01-22 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Insomnia Chronic; Insomnia; Insomnia, Primary; Depression; Depressive Symptoms
Keywords: Metabolism; Metabolomics
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- Waitlist Control (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — Subjects receive 6-8 CBT-I sessions in an individual format.
  Arms: CBT-I

SUMMARY:
This project will examine changes in metabolism and depressive symptoms after receiving CBT-I in 30 subjects with insomnia disorder and MDD.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia Severity Index > 14
* Meet diagnostic criteria for Insomnia
* Meet diagnostic criteria for Major Depressive Disorder
* Either currently taking an SSRI/SNRI or no antidepressant

Exclusion Criteria:

* BMI > 30
* Those with unstable medical conditions defined by change in diagnosis or medication in past 2 months
* Those with clinically significant comorbid psychiatric conditions (e.g., Bipolar disorder)
* Those with known untreated sleep apnea or other clinically significant sleep disorder other than insomnia
* Those currently taking medications that affect sleep or metabolism (e.g., stimulants, thyroid meds)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Metabolomic Assays | Baseline (week 0)
  Blood samples will be collected at enrollment . We will use NMR Spectroscopy to examine serum metabolite changes in patients with insomnia before and after CBT-I, in comparison with therapy control.
Metabolomic Assays | 2 weeks post-treatment (week 10 on average)
  Blood samples will be collected 2 weeks following the completion of CBT-I to examine metabolic markers of response to CBT-I. We will use NMR Spectroscopy to examine serum metabolite changes in patients with insomnia before and after CBT-I, in comparison with therapy control.
Insomnia Severity Index | Baseline (week 0)
  A 7-item (0-4 Likert scale) measure with a total score of 28. The norms for the scale are: 0-7 represents no clinically significant insomnia; 8-14 represents sub-threshold insomnia; 15-21 represents clinical insomnia (moderate severity); 21-28 represents clinical insomnia (severe). The Insomnia Severity Index, the primary outcome of Aim 1, demonstrates good internal consistency (alpha=.74) and is routinely used as the primary outcome measure in insomnia RCTs.
Insomnia Severity Index | 2 weeks post-treatment (week 10 on average)
  A 7-item (0-4 Likert scale) measure with a total score of 28. The norms for the scale are: 0-7 represents no clinically significant insomnia; 8-14 represents sub-threshold insomnia; 15-21 represents clinical insomnia (moderate severity); 21-28 represents clinical insomnia (severe). The Insomnia Severity Index, the primary outcome of Aim 1, demonstrates good internal consistency (alpha=.74) and is routinely used as the primary outcome measure in insomnia RCTs.
Insomnia Severity Index | 3 months post-treatment (week 20 on average)
  A 7-item (0-4 Likert scale) measure with a total score of 28. The norms for the scale are: 0-7 represents no clinically significant insomnia; 8-14 represents sub-threshold insomnia; 15-21 represents clinical insomnia (moderate severity); 21-28 represents clinical insomnia (severe). The Insomnia Severity Index, the primary outcome of Aim 1, demonstrates good internal consistency (alpha=.74) and is routinely used as the primary outcome measure in insomnia RCTs.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No